CLINICAL TRIAL: NCT03334383
Title: Randomized Controlled Trial to Evaluate the Effect of a Retractor Sponge in Postoperative Hospital Stay in Laparoscopic Colorectal Surgery in Patients With Malignancy
Brief Title: Trial for Retractor Sponge Evaluation in Laparoscopic Colorectal Surgery
Acronym: SPONGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, dr. A.B. Smits, Dr. A.M. Smits, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 49877; 49877 (Registry Identifier: CCMO (toetsingonline.nl): ABR form)
Record Dates: First submitted 2017-05-04; First posted 2017-11-07 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Colon Carcinoma; Rectum Carcinoma
Keywords: Laparoscopic colorectal surgery; Retractor sponge; Trendelenburg position; Postoperative complications
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sponge group (Experimental): Patients offered surgery with the retractor sponge
  Interventions: Device: Sponge
- Control group (No Intervention): Patients receiving standard care: surgery in Trendelenburg position

INTERVENTIONS:
Device: Sponge — Compressed cellulose sponge for use in laparoscopic surgery to retract the intestines from the surgical field.
  Other Names: Endoractor, Kawamoto corporation (Osaka, Japan)
  Arms: Sponge group

SUMMARY:
Laparoscopic surgery of the distal colon and rectum requires surgery with an appropriate field of view. A commonly used technique to create a clear exposure is the steep Trendelenburg position in which the patient is positioned in an angle of 15 to 40 degrees with the head down using the effect of gravity to retract the small intestine. This method is associated with haemostatic changes caused by the cranial shift of abdominal organs and blood. Recently, a cellulose compressed sponge was developed as intraoperative retractor, with the aim to keep the small intestines aside while the patient remains in a horizontal position. The safety of the sponge is secured with CE marking. The retractor sponge ensures a clear surgical field and potentially prevents haemostatic instability by avoiding Trendelenburg position. A pilot study in the St Antonius Hospital Nieuwegein has shown that use of the sponge might be associated with shorter hospital stay.

DETAILED DESCRIPTION:
Objective: We study the efficacy of the retractor sponge in laparoscopic colorectal surgery to reduce hospital stay in patients operated for a malignancy. Secondary objectives are duration of surgery, blood-loss, use of diuretics as volume therapy (during surgery as wells as during total hospital stay), postoperative hypoxemia and peri- and postoperative complications.

Study design: Randomized controlled trial, nested within a prospective cohort according to the 'cohort multiple randomized controlled trial' (cmRCT) design.

Study population: Patients with colorectal cancer who undergo laparoscopic surgery, and who have given informed consent to be offered experimental interventions within the PICNIC project. Patient who require open surgery or patients with benign colorectal diseases are excluded for this study.

Intervention: Intraoperative use of the retractor sponge versus usual care, i.e. the Trendelenburg position.

Main study parameters/endpoints: The primary endpoint is length of hospital stay. Secondary endpoints are duration of surgery, blood-loss, use of diuretics (during surgery as wells as during total hospital stay), postoperative hypoxemia and peri- and postoperative surgical, pulmonary and cardiac complications.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The study will be conducted according to the cohort multiple Randomized Controlled Trial (cmRCT) design. Within the PICNIC cohort, we will identify all patients who are eligible for the experimental intervention (use of the sponge) and who have given informed consent to be invited for future experimental interventions. From this sub cohort, we will randomly select a group of patients to whom we will offer surgery with use of the retractor sponge, which they can accept or decline. Eligible patients from the sub cohort who were not randomly selected will undergo standard treatment, i.e. surgery in Trendelenburg position. We do not expect adverse events in patients in the intervention arm, besides dysfunction of the sponge, after which conversion to standard treatment (Trendelenburg position) needs to take place.

ELIGIBILITY:
Inclusion criteria:

* Participant in the PICNIC project (METC 12-510)
* Informed consent obtained for being offered experimental interventions within the PICNIC project
* Informed consent obtained for questionnaires on patient reported outcomes within the PICNIC project
* Planned for laparoscopic surgery of distal colorectal cancer in St. Antonius Hospital

Exclusion Criteria:

* Planned for open colorectal surgery
* Surgery for benign colorectal diseases
* Emergency colorectal surgery
* Inadequate understanding of the Dutch language in speech and/or writing

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative hospital stay (days) | Up to 4 weeks
  Based on a discharge checklist

SECONDARY OUTCOMES:
Operation time | Up to 4 hours
  minutes
Blood-loss peroperative | During surgery time
  ml
Diuretics peroperative and postoperative | Up to 4 weeks (during hospital stay)
  mg
Postoperative hypoxemia | Up to 1 week
  O2 saturation
Peri- and postoperative surgical complications | Up to 4 weeks
  number
Pulmonary complications. | Up to 4 weeks
  number
Cardiac complications | Up to 4 weeks
  number

CONTACTS AND LOCATIONS:
Overall Officials: Anke B Smits, MD, Principal Investigator — St. Antonius Hospital
Locations (1):
- St. Antonius Hospital, Nieuwegein, Utrecht, Netherlands